CLINICAL TRIAL: NCT02188745
Title: Phase II Pre-emptive OsciLLation of ER activitY Levels Through Alternation of Estradiol/Anti-estrogen Therapies Prior to Disease Progression in ER+/HER2- Metastatic or Advanced Breast Cancer
Brief Title: ER Reactivation Therapy for Breast Cancer
Acronym: POLLY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Mary D Chamberlin, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D14122
Record Dates: First submitted 2014-06-24; First posted 2014-07-14 (Estimated); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic; locally advanced; ER+; Estrogen therapy; Estradiol therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Aromatase Inhibitors; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alternating Therapy (Experimental): Study will use an 8-week/16-week alternating regimen of 17B-estradiol/AI (aromatase inhibitor) therapy. Use of only one Aromatase inhibitor throughout the study is preferred.
  17B-estradiol: One tablet containing 2 mg 17B-estradiol will be taken orally three times daily, for a total dose of 6 mg/day.
  Letrozole: One tablet containing 2.5 mg letrozole will be taken orally once per day.
  Anastrozole: One tablet containing 1 mg anastrozole will be taken orally once per day.
  Exemestane: One tablet containing 25 mg exemestane will be taken orally once per day.
  Interventions: Drug: 17B-estradiol; Drug: Letrozole; Drug: Anastrozole; Drug: Exemestane

INTERVENTIONS:
Drug: 17B-estradiol — Anti-estrogen
  Other Names: aromatase inhibitor
Drug: Letrozole — Aromatase inhibitors work by blocking estrogen receptors; they stop a key enzyme (called aromatase) from changing other hormones into estrogen. This lowers estrogen levels in the body, taking away the fuel that estrogen receptor-positive breast cancers need to grow.
  Other Names: Letrozole (Aromatase inhibitor)
Drug: Anastrozole — Aromatase inhibitors work differently from tamoxifen and raloxifene. Instead of blocking the estrogen receptors, they stop a key enzyme (called aromatase) from changing other hormones into estrogen. This lowers estrogen levels in the body, taking away the fuel that estrogen receptor-positive breast cancers need to grow.
  Other Names: Aromatase inhibitor
Drug: Exemestane — Aromatase inhibitors work differently from tamoxifen and raloxifene. Instead of blocking the estrogen receptors, they stop a key enzyme (called aromatase) from changing other hormones into estrogen. This lowers estrogen levels in the body, taking away the fuel that estrogen receptor-positive breast cancers need to grow.
  Other Names: Aromatase inhibitor

SUMMARY:
Before anti-estrogens such as tamoxifen were developed to treat estrogen receptor (ER)-positive breast cancer, high-dose estrogen therapies were used. This seems counterintuitive since anti-estrogens block ER function, while estrogens increase ER function, but these therapies are effective to similar extents for the treatment of metastatic ER+ breast cancer. Estrogen therapies are most effective against cancers that develop resistance to anti-estrogens, likely because such cancers have adapted to grow without ER function, and restoring ER function (with estrogen) is damaging to the cancer cells. In some patients with ER+ breast cancer that becomes resistant to anti-estrogens, treatment with the estrogen 17B-estradiol induces tumor response. Furthermore, when 17B-estradiol-sensitive tumors eventually become resistant to 17B-estradiol, switching back to anti-estrogen therapy is often effective. These observations suggest that cancers can alternate between anti-estrogen-sensitive and 17B-estradiol-sensitive states. The investigators hypothesize that treatment with alternating 17B-estradiol / anti-estrogen therapies on a defined 8-week / 16-week schedule will more effectively prevent cancer growth than continuous treatment with either type of therapy in patients with metastatic anti-estrogen-resistant ER+ breast cancer.

DETAILED DESCRIPTION:
Metastatic breast cancer is rarely cured by current therapies. ER+ breast cancers ultimately become resistant to all available anti-estrogens. Response rates to estrogens are similar to those of anti-estrogens in the metastatic setting. Given that ER+ breast cancers are often responsive to anti-estrogens and estrogens, alternating anti-estrogen/estrogen therapies may be more effective than continuous treatment with either type of agent. Anecdotal evidence indicates that such a strategy of alternating therapies is effective in some patients. Preclinical evidence suggests that anti-estrogen-resistant ER+ breast cancers are sensitized to the anti-tumor effects of estrogens. Such cells harbor subpopulations that can ultimately regain the ability to grow in the presence of estrogens, and revert to their anti-estrogen-sensitive state. The investigators will formally test whether alternating 17B-estradiol/anti-estrogen therapies is effective for the management of anti-estrogen-resistant metastatic ER+/HER2- breast cancer, and to identify molecular biomarkers that predict tumor response to 1) 17B-estradiol and 2) alternating 17B-estradiol/anti-estrogen therapies. If successful, this study would present a novel strategy to manage metastatic ER+/HER2- breast cancer by pre-emptively switching therapies prior to disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥18 years of age with clinical stage IV ER+/HER2- breast cancer, or with locally recurrent ER+/HER2- disease not amenable to therapy for curative intent.
2. Patient must have been treated with an anti-estrogen at any time in their disease history. Combination regimens that include an anti-estrogen and any biologic, or targeted therapy, are permitted (e.g., any CDK inhibitor, everolimus, or any other novel biologics), and are considered to be a single hormonal therapy based regimen.

   * Any number of prior lines of anti-estrogen (i.e., hormonal) therapy is permissible.
   * One line of prior chemotherapy for advanced/metastatic disease is permissible.
3. Histologic documentation of ER strongly+/HER2- breast cancer by core needle biopsy, fine needle aspiration, incisional biopsy, or surgical biopsy of ≥1 site(s) of metastatic or locally advanced disease performed as standard of care within the past 4 months for assessment of eligibility for study participation (except as noted below in c/d/e).

   1. ER strongly+ status defined as ER staining by immunohistochemistry in ≥50% of malignant cell nuclei with an intensity ≥2+ on a scale of 0-3+. These criteria are equivalent to an Allred score ≥6.
   2. HER2-negative status is defined as immunohistochemistry score of 0-1+, or with a FISH ratio of <2 if IHC is 2+ or if IHC has not been done (as per ASCO/CAP definitions). In cases of borderline or equivocal HER2 status, eligibility will be determined by the PI.
   3. Archived tumor specimens: Excess tumor tissue must be available for research purposes. This will include tumor tissue sufficient to make ≥10 five-micron sections; more tumor tissue is preferred.

      Freshly acquired tumor specimens: As part of a clinically indicated biopsy procedure, an additional 1-3 cores or tissue fragments will be obtained by core needle or surgical biopsy for research purposes and FFPE.
   4. Patients with bone-only metastatic disease with a history of ER+/HER2- breast cancer are eligible, and bone biopsy is not required, providing their primary cancer is consistent with the above-described ER and HER2 criteria.
   5. Patients with non-bone metastatic disease in whom a safe and accurate biopsy of recurrent/metastatic disease cannot be readily obtained are also eligible, providing their primary cancer is consistent with the above-described ER and HER2 criteria.
4. Patient must be a candidate for treatment with 17B-estradiol and an aromatase inhibitor.
5. If the most recent therapy was in the adjuvant setting, the recurrence-free interval (time from initiation of adjuvant anti-estrogen therapy to clinical evidence of disease recurrence) must have been ≥2 years.

   If the most recent therapy was in the advanced/metastatic setting, the progression-free interval must have been ≥3 months (except in the case of investigational hormonal therapies).
6. Patient must be post-menopausal based on either a history of an oophorectomy, or ≥1 year of amenorrhea. An elevated serum gonadotropin level and estradiol level in the postmenopausal range (as locally defined) can be used to confirm menopausal status in a subject with <1 year of amenorrhea.
7. Baseline radiographic staging, including specifically either PET/CT, or CT (CAP) and bone scan.
8. Patient must be capable and willing to provide informed written consent for study participation.
9. The following laboratory values must be confirmed for eligibility within 28 days prior to initiation of study therapy:

Hematology panel

* hemoglobin > 9 g/dL
* white blood cell (WBC) count (≥ 2,000/uL)
* platelet count ≥ 75,000/uL Serum biochemistry/metabolic panel
* creatinine ≤ 1.5 x upper limits of normal (ULN)
* total bilirubin ≤ 1.5 x upper limits of normal (ULN)
* ALT and AST ≤ 3.0 x upper limits of normal (ULN) For patients with liver metastasis: < 5 x upper limits of normal (ULN)

Exclusion Criteria:

1. Treatment with fulvestrant within 16 weeks prior to study enrollment.
2. Any other concurrent systemic anti-cancer treatments, including conventional chemotherapeutic agents and biological agents, during the study period.

   Anti-resorptive bone therapies (e.g., bisphosphonates, denosumab) are permitted.
3. Any investigational cancer therapy in the last 3 weeks.
4. Known CNS disease, unless clinically stable for ≥ 3 months.
5. History of any of the following:

   * deep venous thrombosis
   * pulmonary embolism
   * stroke
   * acute myocardial infarction
   * congestive heart failure
   * previous malignancy not treated with curative intent, or with an estimated recurrence risk ≥30%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Clinical benefit | 12 Months
  Determine the rate of clinical benefit from alternating 17B-estradiol/aromatase. Clinical benefit is defined as complete response, partial response or stable disease at 24 weeks per RECIST criteria.

SECONDARY OUTCOMES:
Objective response rate | 8 weeks
  Determine the objective response rate of patients treated with 17B-estradiol therapy for 8 weeks. Objective Response is defined as complete response + partial response as per RECIST criteria; the proportion of patients experiencing objective response on 17B-estradiol will be calculated to determine objective response rate.
Progression-free survival | 12 Months
  Determine the progression-free survival from alternating 17B-estradiol/aromatase inhibitor therapy in patients with advanced ER+ breast cancer. Progression-free survival is defined as the time period from the start of a treatment until the time of cancer progression or death from any cause. Cancer progression will be determined as per RECIST criteria.
Adverse event profiles | 12 Months
  Determine the adverse event profiles of 17B-estradiol and aromatase inhibitors in this patient population. Adverse events will be recorded as Grade 1, 2, 3, or 4. Incidences will be compared within patients over time.
Predictive tumor genetic lesions | 12 Months
  Determine whether specific tumor genetic lesions in ESR1 are predictive of response to 17B-estradiol and/or subsequent aromatase inhibitor therapies. The rates of clinical benefit from 17B-estradiol and/or subsequent AI therapy will be compared between patients with tumors with vs. without genetic lesions in ESR1.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Chamberlin, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (3):
- United States (3):
  - Baystate Medical Center, Springfield, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire